CLINICAL TRIAL: NCT04371588
Title: Effect of Perioperative Muscle Relaxant Model on Postoperative Outcomes in Chinese Patients
Brief Title: Perioperative Muscle Relaxant and Postoperative Outcomes
Acronym: POMPO
Status: Completed | Type: Observational
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Professor, Air Force Military Medical University, China
Other Study IDs: XJH-A-20290110
Record Dates: First submitted 2020-04-27; First posted 2020-05-01 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Complications
Keywords: muscle relaxant; general anesthesia; Chinese patient
MeSH Terms: conditions — Postoperative Complications; Muscle Hypotonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deep neuro-muscular blockade
  Interventions: Other: No Response to Train of Four Stimulation
- Moderate neuro-muscular blockade
  Interventions: Other: 1-2 Response to Train of Four Stimulation

INTERVENTIONS:
Other: No Response to Train of Four Stimulation — No response is observed during Train of Four stimulation monitoring during surgery
  Groups: Deep neuro-muscular blockade
Other: 1-2 Response to Train of Four Stimulation — 1 to 2 response is observed during Train of Four stimulation monitoring during surgery
  Groups: Moderate neuro-muscular blockade

SUMMARY:
Muscle relaxant is usually needed for surgery. However, the optimal depth of neuro-muscular blockade is still on debate. Deep neuro-muscular blockade may benefit the patients during surgery, but may increase the risk of residual blockade after surgery. Residual blockade has been reported to increase risk of morbidity. In this study, we tend to observe the postoperative outcomes in patients undergoing abdominal surgery under general anesthesia. And to compare the outcomes in patients received different depth of neuro-muscular blockade.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Body mass <18 kg/m2
* American Society of Anesthesiologists status I-II
* Patients scheduled for elective laparoscopic colorectal or urological surgery
* Patients received general anesthesia and muscle relaxant
* Patients with written informed consent.

Exclusion Criteria:

* Second surgery during the same admission.
* Outpatient surgery
* Retroperitoneal laparoscopic surgery
* Patients scheduled for mechanical ventilation after surgery
* Patients scheduled for muscle relaxant other than rocuronium
* Patients with pregnancy or planned for breeding
* Patients who are involved in other studies

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for laparoscopic surgery are consecutively screened with inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 999 (Actual)
Dates: Start 2018-03-17 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale of pain at rest at 24 hours after surgery | from end of surgery to 24 hours after surgery
  The intensity of pain is reported by the patient by provide a number between 0 and 10. 0 means no pain, and 10 means unbearable pain. Higher score means stronger pain.
Visual Analogue Scale of pain at cough at 24 hours after surgery | from end of surgery to 24 hours after surgery
  The intensity of pain is reported by the patient by provide a number between 0 and 10. 0 means no pain, and 10 means unbearable pain. Higher score means stronger pain.

SECONDARY OUTCOMES:
Incidence of patients suffering pain at 24 hours after surgery | from end of surgery to 24 hours after surgery
Time to flatus | from end of surgery to flatus, on an average of 3 days
Time to extubation of the endotracheal tube | from end of surgery to removal of the endotracheal tube, on an average of 15 minutes
Incidence of major postoperative complications | from end of surgery to discharge from the hospital, on an average of 5 days
  Incidence of major postoperative complications (including myocardial ischemia, pulmonary infection, respiratory failure, brain ischemia)
Satisfaction score of the Surgeon to the condition during surgery | from start of surgery to end of surgery, on an average of 2.5 hours
  The satisfaction of the Surgeon is measured by a scale from 0-10. 0 is for extremely unsatisfied, 10 is for totally satisfied. Higher score means higher satisfaction. The surgeon is asked to give a number between 0 and 10 to describe his satisfaction.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - First hospital of Beijing University, Beijing, Beijing Municipality
  - Xiehe Hospital of Fujian Medical University, Fuzhou, Fujian
  - First Afiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical School, Wuhan, Hubei
  - Xiehe Hospital of Tongji Medical School, Wuhan, Hubei
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Huaxi Hospital, Chengdu, Sichuan
  - General hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - People's Hospital of Jiangsu, Nanjing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madsen MV, Istre O, Staehr-Rye AK, Springborg HH, Rosenberg J, Lund J, Gatke MR. Postoperative shoulder pain after laparoscopic hysterectomy with deep neuromuscular blockade and low-pressure pneumoperitoneum: A randomised controlled trial. Eur J Anaesthesiol. 2016 May;33(5):341-7. doi: 10.1097/EJA.0000000000000360. PMID 26479510
- [Background] Torensma B, Martini CH, Boon M, Olofsen E, In 't Veld B, Liem RS, Knook MT, Swank DJ, Dahan A. Deep Neuromuscular Block Improves Surgical Conditions during Bariatric Surgery and Reduces Postoperative Pain: A Randomized Double Blind Controlled Trial. PLoS One. 2016 Dec 9;11(12):e0167907. doi: 10.1371/journal.pone.0167907. eCollection 2016. PMID 27936214